CLINICAL TRIAL: NCT06782152
Title: AVEIR™ Leadless Pacemaker Registry in Europe and MIddle East Region
Brief Title: AVEIR™ Leadless Pacemaker Registry in Europe and MIddle East Region (PREMIER LEADLESS)
Status: Not yet recruiting | Type: Observational
Sponsor: King Fahad Armed Forces Hospital (Other Government)
Responsible Party: Principal Investigator, Fayez Bokhari, Medical Director - Head of Cardiology, King Fahad Armed Forces Hospital
Other Study IDs: Version A
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Pacing in Adherence With ESC Cardiac Pacing Guidelines
Keywords: Bradycardia; Sick Sinus Syndrome; Pacemaker; AV Block; Vasovagal Syncope; Heart Diseases; Cardiovascular Diseases; Pathologic Proceses; Arrhytmias, Cardiac
MeSH Terms: conditions — Bradycardia; Sick Sinus Syndrome; Atrioventricular Block; Syncope, Vasovagal; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The AVEIR™ Leadless Pacemaker Registry (herein referred to as "PREMIER LEADLESS Registry") is a prospective, multicenter, International, open label observational study designed to evaluate safety and electrical performances of AVEIR™ leadless pacemakers used in real-world clinical practice and to evaluate clinical outcomes and characteristics of patients treated with these leadless devices.

DETAILED DESCRIPTION:
The AVEIR™ Leadless Pacemaker Registry (herein referred to as "PREMIER LEADLESS Registry") is a prospective, multicenter, International, open label observational study designed to evaluate safety and electrical performances of AVEIR™ leadless pacemakers used in real-world clinical practice and to evaluate clinical outcomes and characteristics of patients treated with these leadless devices. The study aims to evaluate safety profile, electrical performances and clinical outcomes in patients indicated for cardiac pacing after they receive Aveir LP systems. The Aveir VR LP system, for ventricular pacing, and the Aveir AR LP system for atrial pacing, and their concomitant use in the dual chamber configuration (Aveir DR LP system), have received the CE mark. The study also aims to understand clinical characteristics of patients receiving AVEIR™ leadless pacemaker devices in real-world clinical practice. The study Investigators will gather data from routine hospital practices and standard-of-care (SOC) procedures administered to patients. All devices used in these procedures are commercially available and already in use in the participating sites. The structure of this document provides a general overview and methodology of the study and a few specific details such as sample size, follow-up procedures, reporting requirements, and definitions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has clinical indication to cardiac pacing in adherence with ESC cardiac pacing guidelines.
2. Subject is ≥ 18 years of age or age of legal consent, whichever age is greater.
3. Subject agrees to return to clinic for the study follow-up visits.
4. Subject has been informed of the nature of the study, agrees to its provisions and has provided a signed written informed consent, approved by IRB/EC.

Exclusion Criteria:

1. Subject is currently participating in another study that may confound the results of this research.
2. Subject has a life expectancy less than 12 months.
3. Subject is pregnant or nursing or planning pregnancy during the study.
4. Subject has anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the study or to comply with the site standard follow-up visits, for example a mechanical tricuspid

   - Page 3 of 4 [DRAFT] - valve prosthesis or vein thrombosis, which could impede the delivery of implantable devices as planned by the implanters.
5. Subject is allergic/hypersensitive to <1 mg dexamethasone sodium phosphate.
6. Subject is implanted with an electrically active implantable medical device with stimulation capabilities at risk to be impacted by the Aveir Link Module telemetry.
7. Subject has known pacemaker syndrome, if that condition, in the investigator's opinion, represents a contraindication to the implant of the planned pacemaker.
8. Subject has pacing induced cardiomyopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject clinically indicated to receive a Leadless Pacemaker in adherence with ESC cardiac pacing guidelines.
Sampling Method: Probability Sample
Enrollment: 1698 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint is 1 year incidence rate of leadless device-related or procedure-related major complications. AveirTM LP systems | 12 momths
  Major complications are defined as events related to the leadless pacing system or leadless pacing system implant procedure resulting in death, permanent loss of device function due to mechanical or electrical dysfunction, hospitalization, prolonged hospitalization by at least 48 h, or system revision AveirTM LP systems
Acceptable ventricular pacing thresholds and R-wave amplitudes measured at 12 months. | 12 months
  Ventricular pacing threshold is considered acceptable if <2.0 V at 0.4 ms and R-wave amplitude is considered acceptable if >5.0 mV or ≥ of the implant value
Acceptable atrial pacing thresholds and P-wave amplitudes as measured at 12 months. | 12 months
  atrial capture threshold is considered acceptable if ≤3.0 V at 0.4 ms and atrial sensing Amplitude is considered adequate if P wave ≥1.0 mV.

SECONDARY OUTCOMES:
Freedom from device- or procedure-related major complications at 24 months | 24 months
  Major complications are defined as events related to the leadless pacing system or leadless pacing system implant procedure resulting in death, permanent loss of device function due to mechanical or electrical dysfunction, hospitalization, prolonged hospitalization by at least 48 h, or system revision.
All adverse events, regardless device- or procedure-relatedness. | 48 months
Implant success rate and reasons for unsuccessful implant. | 24 months
Number of device repositioning at time of implantation. | 24 months
Implant duration, fluoroscopy duration, and time from implant to hospital discharge. | 24 months
Final LP placement site. | 24 months
Demographics and medical history, with specific focus on indication for pacemaker implant and reasons for the choice of leadless pacemakers. | 24 months
Device longevity, as displayed by the programmer at each visit. | 48 months
Device programming and pacing and sensing conditions which may impact longevity. | 48 months
Need for and success of device retrieval. | 48 months
Number of hospitalizations and mortality. | 48 months
Upgrade from Aveir VR to Aveir DR and from Aveir AR to Aveir DR.and Communication i2i success rate. | 48 months
Development of pacing induced cardiomyopathy | 48 months